CLINICAL TRIAL: NCT02826070
Title: Efficacy of Long-term Telbivudine Treatment on Histological Improvements in Patients With Chronic Hepatitis B (EFFORT Further Extension Study)
Brief Title: EFFORT Further Extension Study
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: Major Science and Technology Special Project of China Twelfth-Five-Year Project (Unknown); Novartis (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MOH-09
Record Dates: First submitted 2016-06-27; First posted 2016-07-07 (Estimated); Last update posted 2016-07-07 (Estimated); Status verified 2016-06

CONDITIONS: Hepatitis B, Chronic
Keywords: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Telbivudine; adefovir dipivoxil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Off-treatment (Other): Patients who had stopped treatment during EFFORT extension study could receive 2-year off-treatment follow-up. All the patients in Part I will be followed up at the interval of 12 weeks. For these patients, if they have hepatitis flare during follow-up, they will be re-treated with telbivudine combined with adefovir for the left study period ( the total study period is 2 years) and followed up at the interval of 12 weeks. Hepatitis flare is defined as HBV DNA>4 Log10 copies/mL with either ALT≥5 times upper limit of normal (ULN) or TBIL≥2×ULN，or 2 ≤ALT ≤5 ×ULN (at two consecutive visits at least 2 weeks apart) and total bilirubin (TBIL) <2×ULN.
  Interventions: Other: off-treatment follow-up
- On-treatment (Other): Patients with continuous treatment during EFFORT extension study will continue treatment, without off-treatment rule in the further extension study. The treatment strategy is depended on the HBV DNA level of each individual, that is, for patients with negative HBV DNA level (defined as HBV DNA <20 IU/mL) will continue their previous treatment strategy; and for patients with positive HBV DNA level (defined as HBV DNA>=20 IU/mL) will receive the combination therapy of telbivudine and adefovir, irrespective of their previous treatment strategy. All the patients in Part II will be followed up at the interval of 24 weeks until they complete the 2-year on-treatment follow-up. Patients will be conducted liver biopsy at the sixth year of treatment. All the patients with telbivudine monotherapy will be switched to telbivudine plus adefovir once confirmed HBV DNA breakthrough developed.
  Interventions: Drug: Telbivudine; Drug: Adefovir dipivoxil

INTERVENTIONS:
Drug: Telbivudine — Telbivudine, 600mg, oral, daily
  Arms: On-treatment
Drug: Adefovir dipivoxil — Adefovir dipivoxil 10mg, oral, daily
  Arms: On-treatment
Other: off-treatment follow-up
  Arms: Off-treatment

SUMMARY:
The purpose of this study is to demonstrate that long-term treatment (up to six years) with telbivudine or telbivudine plus adefovir results in the regression in liver inflammation and fibrosis/cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who completed EFFORT extension study.
2. Patients who had baseline (that is the week 0 of EFFORT study) HBV DNA <9 Log copies/mL and ALT ≥2×ULN.
3. Patients who are willing to participate in the further extension study.
4. Patient is willing and able to comply with the study drug regimen and all other study requirements.
5. Patients must give written informed consent before any assessment is performed.

Exclusion Criteria:

1. Poor compliance judged by investigators

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2015-04; Primary Completion 2016-10 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with histological improvement (≥2-point decrease in the Knodell necroinflammatory score and no worsening in Ishak fibrosis score). | Week 48

SECONDARY OUTCOMES:
Percentage of patients achieving hepatitis B virus (HBV) DNA <300copies/mL at week 48 and 96 in on-treatment group | week 48, week 96
Percentage of patients with HBeAg loss or HBeAg seroconversion at week 48 and 96 in on-treatment group | week 48, week 96
Percentage of patients with HBsAg loss or HBsAg seroconversion at week 48 and 96 in on-treatment group | week 48, week 96
The percentage of patients with alanine aminotransferase (ALT) normalization at week 48 and 96 in on-treatment group | week 48, week 96
Percentage of patients with HBV DNA breakthrough at week 48 and 96 in on-treatment group | week 48, week 96
Percentage of patients with genotypic resistance among the patients with HBV DNA breakthrough at week 48 and 96 in on-treatment group | week 48, week 96
Incidence of adverse effect at week 48 and 96 in on-treatment group | week 48, week 96
Percentage of patients with glomerular filtration rate (GFR) shifting to >90 mL/min/1.73 m2 for patients with GFR <90 mL/min/1.73 m2 at baseline of EFFORT study at week 48 and 96 in on-treatment group | week 48, week 96
Sustained response rate of durability of HBeAg seroconversion at week 48 and 96 in off-treatment group | week 48, week 96
Percentage of patients who re-achieved ALT normalization and HBV DNA <300 copies/mL in the patients retreated who developed hepatitis flare after stopping treatment in off-treatment group | week 96
Incidence of abnormal laboratory examination at week 48 and 96 in on-treatment group | week 48, week 96
Percentage of hepatitis flare at week 48 and 96 in off-treatment group | week 48, week 96

CONTACTS AND LOCATIONS:
Overall Officials: Jinlin Hou, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (20):
- China (20):
  - 302 Military Hospital Of China, Beijing, Beijing Municipality
  - Beijing Ditan Hospital, Beijing, Beijing Municipality
  - BeiJing YouAn Hospital ,Capital Medical University, Beijing, Beijing Municipality
  - Department of infectious disease, First Hospital of Peking University, Beijing, Beijing Municipality
  - People's Hospital of Beijing University, Beijing, Beijing Municipality
  - The Second Affiliated of ChongQing University of Medical Science, Chongqing, Chongqing Municipality
  - Department of Infectious Disease, Nanfang Hospital, Guangzhou, Guangdong
  - No. 8 People's Hospital In GuangZhou, Guangzhou, Guangdong
  - The Third Hospital of Sun Yat-Sen University, Guangzhou, Guangdong
  - Tongji Hospital of Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - Xiangya Hospital Central-South Univrsity, Changsha, Hunan
  - No.81 Hospital of PLA, Nanjing, Jiangsu
  - First Hospital .Jilin Unniversity, Changchun, Jilin
  - ShengJing Hospital of China Medical University, Shengyang, Liaoning
  - JiNan Infectious Diseases Hospital, Jinan, Shandong
  - Changhai Hospital affiliated to Second Military Medical University, Shanghai, Shanghai Municipality
  - Huashan Hospital，Fudan University, Shanghai, Shanghai Municipality
  - Shanghai Ruijin Hospital, Shanghai, Shanghai Municipality
  - Tangdu Hospital, XiAn, Shanxi
  - The First Affiliated Hospital of College of Medicine, Zhejiang University, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided